CLINICAL TRIAL: NCT02247453
Title: Plasma microRNA Profiling as First Line Screening Test for Lung Cancer Detection: a Prospective Study
Acronym: BIOMILD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Ugo Pastorino, MD, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: INT11-21
Record Dates: First submitted 2014-04-24; First posted 2014-09-25 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer
Keywords: lung cancer; clinical trial; screening; microRNA; biomarkers
MeSH Terms: conditions — Lung Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Screening (Experimental): Healthy heavy smokers aged 50-75 years
  Interventions: Other: screening

INTERVENTIONS:
Other: screening — All subjects undergo baseline LDCT examination, spirometry and miRNA profiling. Individuals with negative miRNA profile repeat the plasma assay at 3 years. Individuals with low-risk miRNA profile repeat the plasma assay and LDCT at 2 years, without additional diagnostic examinations if not required by the screening protocol.
  Individuals with high-risk miRNA profile undergo additional diagnostic examinations consisting in PET in case of concurrent suspicious or positive CT, or WB MRI +- needle aspiration biopsy in case of negative CT.

SUMMARY:
In the present project we propose a large prospective study in heavy smokers volunteers based on plasma miRNA profiling to assess its efficacy as a first line screening test for lung cancer detection.

The study will be articulated in different phases: i) analysis of 1000 plasma samples of disease-free smokers already collected in our biological repository in the last two years ii) de-novo enrollment of 4000 smoking volunteers, collection of their blood samples and inclusion in a program of active surveillance on the basis of their miRNA risk profile iii) assessment of miRNA expression profile using a custom made microfluidic card containing the 24 miRNA previously identified in the diagnostic signatures iii) bioinformatic analyses of miRNA ratios in the cohort in order to determine which individuals are in presence or will develop lung cancer and in particular the aggressive form of the disease iv) assessment of the best diagnostic and treatment algorithm for subjects with suspicious miRNA profiles v) functional validation of miRNAs as novel therapeutic targets using novel cellular genetically engineered models of transformation and patients' tumorgrafts models.

DETAILED DESCRIPTION:
Three decades of research have shown that radiological screening of heavy smokers can detect resectable early lung cancers with higher frequency but benefit on mortality is still debated. The preliminary results of the first two randomized spiral-CT screening trials appear conflicting, with one study showing no benefit and the other a limited mortality reduction (-7%). In the next 3-4 years the ongoing randomised trials in Europe will provide conclusive data on the efficacy of CT-screening for lung cancer. Nonetheless, no major impact on mortality is to be expected.

A possible explanation of these finding is that not all aggressive lung tumors arise from identifiable slow-growing precursors, thus suggesting a possible paradigm shift in our understanding of the natural history of lung cancer. In this respect the identification of biologic and molecular features of indolent and aggressive disease could be useful to define clinical predictors of high risk lesions and select suitable cohorts of patients who might benefit of current treatments as well as to identify genetic signatures that might represent novel therapeutic targets.

The investigators recently reported that microRNA (miRNA) expression expression profiles in tumors and, for the first time, also in normal lung tissue are indicative of aggressive lung cancer development and, of remarkable interest, that specific miRNA signatures can be identified in plasma samples of patients up to two years before spiral-CT detection of the disease, and able to identify the occurrence of early metastatic but spiral-CT invisible lung tumors or small spiral-CT detected lesions with aggressive potential.

In the present project we propose a large prospective study in heavy smokers volunteers based on plasma miRNA profiling to assess its efficacy as a first line screening test for lung cancer detection.

The study will be articulated in different phases: i) analysis of 1000 plasma samples of disease-free smokers already collected in our biological repository in the last two years ii) de-novo enrollment of 4000 smoking volunteers, collection of their blood samples and inclusion in a program of active surveillance on the basis of their miRNA risk profile iii) assessment of miRNA expression profile using a custom made microfluidic card containing the 24 miRNA previously identified in the diagnostic signatures iii) bioinformatic analyses of miRNA ratios in the cohort in order to determine which individuals are in presence or will develop lung cancer and in particular the aggressive form of the disease iv) assessment of the best diagnostic and treatment algorithm for subjects with suspicious miRNA profiles v) functional validation of miRNAs as novel therapeutic targets using novel cellular genetically engineered models of transformation and patients' tumorgrafts models.

Overall, the results of this large prospective study will permit to establish the potential of our plasma microRNA assay as a first-line screening test for lung cancer detection in a routine clinical practice for high-risk population screening with a low cost, non toxic and non invasive procedure. Moreover, the related functional studies foreseen in the project could lead to the identification of novel, miRNA targeted, therapeutic approaches for this malignancy.

ELIGIBILITY:
Inclusion Criteria:

* current heavy smokers of ≥ 30 pack/years, aged 50-75, or former smokers with the same smoking habits having stopped from 10 years or less;
* current or former smokers of < 30 pack/years, aged ≥ 50, with additional risk factors such as family history of lung cancer, prior diagnosis of chronic obstructive pulmonary disease (COPD) or pneumonia, professional exposure to known carcinogens (i.e. asbestos).

Exclusion Criteria:

* subjects with neoplasms within previous five years-
* subjects with suspected lung nodules under investigation

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4119 (Actual)
Dates: Start 2013-01; Primary Completion 2019-11 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Reduction of false positive cases in lung cancer detection in heavy smokers volunteers through plasma miRNA profiling as a first line screening test | 3 years

SECONDARY OUTCOMES:
overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ugo Pastorino, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boeri M, Verri C, Conte D, Roz L, Modena P, Facchinetti F, Calabro E, Croce CM, Pastorino U, Sozzi G. MicroRNA signatures in tissues and plasma predict development and prognosis of computed tomography detected lung cancer. Proc Natl Acad Sci U S A. 2011 Mar 1;108(9):3713-8. doi: 10.1073/pnas.1100048108. Epub 2011 Feb 7. PMID 21300873
- [Background] Sozzi G, Pastorino U, Croce CM. MicroRNAs and lung cancer: from markers to targets. Cell Cycle. 2011 Jul 1;10(13):2045-6. doi: 10.4161/cc.10.13.15712. No abstract available. PMID 21623159
- [Background] Pastorino U, Rossi M, Rosato V, Marchiano A, Sverzellati N, Morosi C, Fabbri A, Galeone C, Negri E, Sozzi G, Pelosi G, La Vecchia C. Annual or biennial CT screening versus observation in heavy smokers: 5-year results of the MILD trial. Eur J Cancer Prev. 2012 May;21(3):308-15. doi: 10.1097/CEJ.0b013e328351e1b6. PMID 22465911
- [Background] Boeri M, Pastorino U, Sozzi G. Role of microRNAs in lung cancer: microRNA signatures in cancer prognosis. Cancer J. 2012 May-Jun;18(3):268-74. doi: 10.1097/PPO.0b013e318258b743. PMID 22647364
- [Background] Pastorino U. Current status of lung cancer screening. Thorac Surg Clin. 2013 May;23(2):129-40. doi: 10.1016/j.thorsurg.2013.01.018. PMID 23566965
- [Background] Pastorino U, Sverzellati N. Lung cancer: CT screening for lung cancer--do we have an answer? Nat Rev Clin Oncol. 2013 Dec;10(12):672-3. doi: 10.1038/nrclinonc.2013.198. Epub 2013 Nov 5. No abstract available. PMID 24189470
- [Background] Sozzi G, Boeri M, Rossi M, Verri C, Suatoni P, Bravi F, Roz L, Conte D, Grassi M, Sverzellati N, Marchiano A, Negri E, La Vecchia C, Pastorino U. Clinical utility of a plasma-based miRNA signature classifier within computed tomography lung cancer screening: a correlative MILD trial study. J Clin Oncol. 2014 Mar 10;32(8):768-73. doi: 10.1200/JCO.2013.50.4357. Epub 2014 Jan 13. PMID 24419137
- [Background] Fortunato O, Boeri M, Verri C, Conte D, Mensah M, Suatoni P, Pastorino U, Sozzi G. Assessment of circulating microRNAs in plasma of lung cancer patients. Molecules. 2014 Mar 10;19(3):3038-54. doi: 10.3390/molecules19033038. PMID 24619302
- [Background] Sestini S, Boeri M, Marchiano A, Pelosi G, Galeone C, Verri C, Suatoni P, Sverzellati N, La Vecchia C, Sozzi G, Pastorino U. Circulating microRNA signature as liquid-biopsy to monitor lung cancer in low-dose computed tomography screening. Oncotarget. 2015 Oct 20;6(32):32868-77. doi: 10.18632/oncotarget.5210. PMID 26451608
- [Background] Boeri M, Sestini S, Fortunato O, Verri C, Suatoni P, Pastorino U, Sozzi G. Recent advances of microRNA-based molecular diagnostics to reduce false-positive lung cancer imaging. Expert Rev Mol Diagn. 2015 Jun;15(6):801-13. doi: 10.1586/14737159.2015.1041377. Epub 2015 Apr 30. PMID 25924864
- [Derived] Boeri M, Sabia F, Ledda RE, Balbi M, Suatoni P, Segale M, Zanghi A, Cantarutti A, Rolli L, Valsecchi C, Corrao G, Marchiano A, Pastorino U, Sozzi G. Blood microRNA testing in participants with suspicious low-dose CT findings: follow-up of the BioMILD lung cancer screening trial. Lancet Reg Health Eur. 2024 Sep 16;46:101070. doi: 10.1016/j.lanepe.2024.101070. eCollection 2024 Nov. PMID 39319217
- [Derived] Zyla J, Dziadziuszko R, Marczyk M, Sitkiewicz M, Szczepanowska M, Bottoni E, Veronesi G, Rzyman W, Polanska J, Widlak P. miR-122 and miR-21 are Stable Components of miRNA Signatures of Early Lung Cancer after Validation in Three Independent Cohorts. J Mol Diagn. 2024 Jan;26(1):37-48. doi: 10.1016/j.jmoldx.2023.09.010. Epub 2023 Oct 20. PMID 37865291
- See also: clinical trial website — http://www.biomild.org